CLINICAL TRIAL: NCT02434627
Title: Sodium Nitrate for Muscular Dystrophy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro35228
Record Dates: First submitted 2015-04-28; First posted 2015-05-05 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2016-10

CONDITIONS: Becker Muscular Dystrophy
Keywords: Becker; Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — sodium nitrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sodium Nitrate (Beetroot Juice) (Experimental): Sodium nitrate in the form of beetroot juice will be administered orally. Patients will be assessed with a number of functional muscle assessments.
  Interventions: Drug: Sodium Nitrate

INTERVENTIONS:
Drug: Sodium Nitrate — Patients will be given sodium nitrate daily in the form of beetroot juice.

SUMMARY:
The investigators' previous work in males with Becker Muscular Dystrophy shows that functional sympatholysis is restored by acute inorganic nitrate supplementation. This was translated from work using the mdx mouse model of dystrophinopathy. Recent work has shown that there is a frank improvement in grip strength when mdx mice are treated with an inorganic Nitric Oxide (NO) donor. The purpose of this study is to determine if chronic treatment with an inorganic NO donor can benefit patients with muscular dystrophy beyond blood flow regulation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of muscular dystrophy
* Age 15-45 years of age
* Ambulatory
* No clinical evidence of heart failure
* Maximum voluntary contraction, measured by hand grip dynamometer, of 20-40 kg

Exclusion Criteria:

* Hypertension, diabetes, or heart failure by standard clinical criteria
* Elevated B-type Natruiretic Peptide level (>100 pg/ml)
* Left Ventricular Ejection Fraction < 50%
* Wheelchair bound
* Cardiac rhythm disorder, specifically: rhythm other than sinus, Supraventricular Tachycardia, atrial fibrillation, ventricular tachycardia
* Continuous ventilatory support
* Liver disease
* Renal impairment
* Contraindications to NO donors (use of nitrates, alpha-blockers, CYP3A inhibitors, amlodipine, or Phosphodiesterase type 5 (PDE5) inhibitors) Glucocorticoid therapy and prophylactic use of Angiotensin Converting Enzyme (ACE) inhibitors and beta-blockers for cardiac protection will not be exclusion criteria.
* Maximum voluntary contraction of less than 20 kg or greater than 40 kg
* Ventilation Devices (Continuous Positive Airway Pressure (CPAP), Bilevel Positive Airway Pressure (BiPAP))

Ages: 15 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2015-06; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Change in maximal handgrip strength | Change from baseline in handgrip strength at 3 months

SECONDARY OUTCOMES:
Change in muscle function - Performance of Upper Limb Scale | Change from baseline in muscle function - the Performance of Upper Limb Scale at 3 months
  Change in functional muscle assessment as measured by the Performance of Upper Limb Scale
Change in muscle tissue markers - histology and proteomics | Change from baseline in muscle tissue markers at 3 monthss
  Change in tissue markers such as neuronal Nitric Oxide Synthase (nNOS) content and location and nitrosative stress by histology and proteomics
Change in systolic wall strain - imaging | Change from baseline in cardiac systolic wall strain at 3 months
  Change in the cardiac wall strain as measured by Cardiac Magnetic Resonance Imaging
Change in muscle function - North Star Ambulatory Assessment | Change from baseline in muscle function - North Star Ambulatory Assessment at 3 months
  Change in functional muscle assessment as measured by the North Star Ambulatory Assessment
Change in muscle function - 6 minute walk test | Change from baseline in muscle function - 6 minute walk test at 3 months
  Change in functional muscle assessment as measured by the 6 minute walk test

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Victor, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No